CLINICAL TRIAL: NCT03657914
Title: A Multi-center Clinical Study on the Feasibility and Safety of Radical Resection of Single-hole Inflatable Mediastinal Mirror Synchronization With Laparoscopic Esophageal Carcinoma
Brief Title: Radical Resection of Single-hole Inflatable Mediastinal Mirror Synchronization With Laparoscopic Esophageal Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qingdong Cao (Other)
Responsible Party: Sponsor-Investigator, Qingdong Cao, Director of Thoracic and Cardiovascular Surgery Department, Fifth Affiliated Hospital, Sun Yat-Sen University
Organization: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDWY.XXW.001
Record Dates: First submitted 2018-08-06; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Esophagus Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inflatable mediastinal mirror (Experimental): Patients with especially esophageal squamous cell carcinoma ( ESCC ) who meet the inclusion criteria and do not meet the exclusion criteria will undergo radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma, and will be followed up until 3 years after discharging from the hospital.
  Interventions: Procedure: Single-hole inflatable mediastinal mirror

INTERVENTIONS:
Procedure: Single-hole inflatable mediastinal mirror — The radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma is new minimally invasive operation for esophageal carcinoma. All enrolled subjects will receive this operation for their ESCC.

SUMMARY:
This study is evaluating the feasibility and safety of radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma, as well as the clinical value of the radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma as a new minimally invasive operation for esophageal carcinoma.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open clinical study in which 155 patients (including 5% shedding rate) who require surgical treatment are scheduled to be included in the study. Prior to any screening process, each subject / legal guardian should sign the informed consent form. Screening tests are used to determine whether each subject is eligible for the study. Eligible subjects who meet the standard will be treated with radical resection of single-hole inflatable mediastinal mirror synchronization with laparoscopic esophageal carcinoma and followed up until 3 years postoperatively. Primary study outcome are the prioperative complication rate and the number of intraoperative lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85 years male and female
* Patients with esophageal squamous cell carcinoma diagnosed by cytological or histological examination, requires surgical treatment
* Patients in tumor stage of T1-2N0-1M0 confirmed by ultrasonic gastroscopy preoperatively;Or patients in T3N1M0 (IIIa) reached PR after neoadjuvant radio(chemo-) therapy, suitable for surgical resection
* The tumor located in the chest or abdomen segment of esophagus
* No surrounding vital organs were invaded and no distant metastasis
* No obvious enlargement was shown in supraclavicular and retroperitoneal lymph nodes, no evidence of distant metastasis (M0)
* Vital organs function normally: lung functions normally and could stand general anesthesia; NYHA heart function grade 0 ~ 1
* Informed consent was signed as voluntarily before study, and patients and/or the legal representatives have the ability to fully understand test content/result, process and possible adverse reactions, and patients could comply with the requirements of the follow-up scheme
* Reproductive women must show a negative pregnancy test, and it should be confirmed that both the women patient and her spouse are taking contraceptives recognized by researchers, and should keep taking this contraceptive by signing the informed consent until 3 months after the study was finished.

Exclusion Criteria:

* Patients with other malignant tumors at the same time
* Patients having surgery history of esophageal or gastric resection
* Patients having a history of mediastinal surgery or vast peritoneal adhesion
* Patients with heart thromboembolism at the same time
* People with psychological, mental or nervous system diseases
* Cachexia, severe malnutrition patients
* Patients with history of recent recurrence of gastric ulcer, stomach bleeding and other severe basic diseases
* Patients with blood coagulation dysfunction, HIV antibody positive, or surgical contraindications such as clinically poorly controlled serious infection
* The subjects with other associated disease (such as liver and renal dysplasia, etc.) or drug combination, which could influence the study results recognized by the researchers
* Patients participating in another clinical study
* Patients with surgical instruments material allergy, or allergic constitution
* The subjects are not judged by investigator to participate in this Clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Perioperative complication rate | Through operation completion, an average of 12 days
  Perioperative complications include: pulmonary infection, respiratory failure, managed pleural effusion, heart failure, myocardial infarction, managed arrhythmia, anastomotic fistula or gastric fistula, recurrent laryngeal nerve injury, chylothorax, unscheduled reoperation
Number of lymph nodes dissected | During the operation
  number of lymph nodes dissected during operation

SECONDARY OUTCOMES:
Intraoperative bleeding volume | During the operation
  Calculation of intraoperative bleeding with ml/kg
Operative time | During the operation
  Calculate the operating time in minutes
Proportion of patients undergoing thoracotomy or laparotomy | During the operation
  The ratio of the number of patients converted to thoracotomy or laparotomy to the total number of patients undergoing surgery
Intraoperative mortality | During the operation
  The ratio of the number of patients who died during the operation to the number of patients who underwent the operation
Postoperative hospital stay | Up to 2 weeks after the operation
  The days of postoperative hospitalization
Postoperative pain score | 1-3 days after the operation
  Daily pain scores were recorded by VAS (Visual Analogue Scale/Score) 1-3 days after operation
Postoperative icu monitoring time | 0-12 days after the operation
  If the patient needs to be transferred to ICU after operation, stay in icu monitoring time should be observed
Incidence of adverse events during and after operation | 3 years
  Special attention is paid to observing whether arrhythmias need to be dealt with during the operation (record the types of arrhythmias, treatment methods, medication, time of occurrence, possible causes)
Postoperative drainage | 0-12 days after the operation
  Total postoperative thoracic or mediastinal drainage (ml/kg)
Postoperative drainage tube indwelling time | 0-12 days after the operation
  The retention time of different types of drainage tube

OTHER OUTCOMES:
Local recurrence rate of tumor within 3 years | 3 years
  The rate of tumor recurrence or metastasis

CONTACTS AND LOCATIONS:
Overall Officials: Liu Shaoxuan, master, Study Chair — Office of clinical research center
Locations (21):
- China (21):
  - Beijing Chao-yang Hospital, Beijing, Beijing Municipality
  - Affiliated Daping Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - Xiangyang No.1 People's Hospital, Xiangyang, Hubei
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiansu Cancer Hospital, Nanjing, Jiangsu
  - Jining No.1 People's Hospital, Jining, Shandong
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - General Hospital of Ningxia Medical University, Yinchuan, The Ningxia Hui Autonomous Region
  - Affiliated Tumor Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang